CLINICAL TRIAL: NCT05474053
Title: Testing P2Y12 Platelet Inhibitors Generics Beyond Bioequivalence: A Parallel Single-blinded Randomized Trial
Brief Title: Testing P2Y12 Platelet Inhibitors Generics Beyond Bioequivalence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Said, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: tica trial
Record Dates: First submitted 2022-07-19; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Cardiovascular Diseases; Acute Coronary Syndrome
MeSH Terms: conditions — Cardiovascular Diseases; Acute Coronary Syndrome | interventions — Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The volunteers were randomly allocated to 2 groups, one receiving the brand drug and the other receiving the generic, each receiving a code indicating his/her group and the key of the codes could only be revealed by the principal investigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brilique group (Experimental): volunteers in the Brilique group received a loading dose of 180 mg brand Brilique® (AstraZeneca , Sweden) then 90 mg twice daily regimen for 4 days
  Interventions: Drug: Ticagrelor 90mg (Brilique)
- Ticaloguard group (Experimental): volunteers in the Ticaloguard group received the Egyptian made generic ticalogaurd in a loading dose of 180 mg then 90 mg twice daily regimen for 4 day
  Interventions: Drug: Ticagrelor 90mg (Ticaloguard)

INTERVENTIONS:
Drug: Ticagrelor 90mg (Brilique) — compare the efficacy and safety of ticagrelor generically named Ticaloguard® compared to its brand Brilique® in healthy volunteers
  Other Names: Brilique
  Arms: Brilique group
Drug: Ticagrelor 90mg (Ticaloguard) — compare the efficacy and safety of ticagrelor generically named Ticaloguard® compared to its brand Brilique® in healthy volunteers
  Arms: Ticaloguard group

SUMMARY:
This is a pilot study that was conducted to prove the efficacy and safety of ticagrelor generically named Ticaloguard® compared to its brand Brilique® in healthy volunteers. we advocate comparing the clinical efficacy rather than simple bioequivalence comparison.

DETAILED DESCRIPTION:
Cardiovascular diseases are the leading cause of death worldwide. Ticagrelor, is an oral antiplatelet drug used in acute coronary syndrome. Although generic drugs are approved for their bioequivalence to the original product, they are not necessarily to be therapeutically equivalent. This study was conducted to prove the efficacy and safety of ticagrelor generically named Ticaloguard® compared to its brand Brilique® in healthy volunteers. A loading dose of 180 mg ticagrelor named Brilique® or Ticaloguard® followed by a 90 mg twice daily regimen as maintenance dose was given to 14 and 15 volunteers in Ticaloguard and Brilique groups, respectively. The platelet aggregation on adenosine diphosphate (ADP) agonist was assessed at different time intervals .

ELIGIBILITY:
Inclusion Criteria:

volunteers of both sexes, aged between 18-64 years old

Exclusion Criteria:

* volunteers with any abnormalities in the complete blood count (CBC) at entry time
* those with any medical conditions contraindicated with antiplatelet therapy
* those taking aspirin, non-steroidal anti-inflammatory drugs (NSAIDs), or any over the counter medications (OTC) that contain medication such as, antihistamines, antibiotics in the previous month
* volunteers with history of blood disorders or bleeding diathesis.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2021-11-13 (Actual); Primary Completion 2021-11-28 (Actual); Study Completion 2021-11-28 (Actual)

PRIMARY OUTCOMES:
testing degree of platelet inhibition of Ticalouguard versus the brand Brilique | 1 month
  Testing the degree of platelet inhibition in both groups through performing platelet aggregation testing using Adenosine diphosphate as agonist

CONTACTS AND LOCATIONS:
Overall Officials: Nirmeen sabry, MD, Study Director — Faculty of pharmacy, Cairo university
Locations (1):
- Faculty of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No